CLINICAL TRIAL: NCT02870751
Title: Developing A Human Challenge Model For Evaluating Vaccines Against ST-producing Enterotoxigenic Escherichia Coli
Brief Title: Human Challenge Model With ST-only Enterotoxigenic Escherichia Coli
Acronym: ETECvacWP2
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bergen (Other)
Collaborators: University of Maryland (Other); Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Kurt Hanevik, PostDoc, Principal investigator, University of Bergen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NRC234364
Record Dates: First submitted 2016-08-13; First posted 2016-08-17 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Diarrhea, Infantile
Keywords: ETEC; human challenge study; heat stable toxin; tourist diarrhea; diarrhea; enterotoxigenic
MeSH Terms: conditions — Diarrhea, Infantile; Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ST-only ETEC strain TW11681 or TW10722 (Experimental): Oral inoculum of several doses of bacteria to establish range to achieve diarrhea attack rate in around 70% of volunteers.
  Interventions: Biological: TW11681 or TW10722

INTERVENTIONS:
Biological: TW11681 or TW10722

SUMMARY:
Heat stable toxin (ST) producing ETEC strains are important causes of childhood diarrhea in many countries. Vaccine candidates targeting ST are in development. A human challenge model using an epidemiologically relevant enterotoxigenic E.coli (ETEC) strain expressing ST, but not other diarrhea inducing toxins like heat labile toxin (LT), is necessary to perform an early and efficient evaluation of an ST-toxoid based vaccine.

In this controlled human infection study the investigators will assess the safety of a ST-only producing ETEC strain and the dose needed to achieve an attack rate of 70% in healthy human volunteers.

DETAILED DESCRIPTION:
The investigators have evaluated the ST-only ETEC strain TW10722 in volunteers previously, and will also evaluate the ETEC strain TW11681, an ETEC family 8, serotype O19:H45, expressing STh, CFA/I, and CS21. These strains have been selected because it is a good representative of one of the most important ETEC families commonly associated with childhood ETEC diarrhea. The TW10722 will also be evaluated at higher dose if TW11681 does not work well.

After screening including routine blood sampling, intestinal lavage and pre-challenge sampling will be done. Volunteers will then be admitted three at a time to Haukeland University Hospital and isolated before receiving the oral bacterial inoculum doses, starting with 10^6 and increasing one log per round until a safe dose that elicits diarrhoea is found. Fine adjustment of the dose needed for a diarrhea attack rate of 70% will then be done in the remaining volunteers. Volunteers will be monitored for a range of symptoms, stool output and adverse events.

Antibiotic treatment will be administered at certain predetermined severities of diarrheal disease, or after 5 days to eradicate the ETEC infection in all volunteers before leaving the hospital. Volunteers will be monitored and sampled again at day 10, 28 and 365 after infection. Serum, plasma, stool, intestinal lavage and PBMC samples will be obtained before, during and after the ETEC infection to evaluate immune responses and potential correlates of protection.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent before initiation of any study procedures.
* Healthy as judged by the Principal Investigator (PI) and determined by medical history, physical examination, and medication history.
* Within 15 days of vaccination, have normal screening laboratories for white blood cells (WBC), hemoglobin (Hgb), platelets, absolute neutrophil count (ANC), sodium, potassium, chloride, bicarbonate, blood urea nitrogen (BUN), creatinine, alanine aminotransferase (ALT), C-reactive protein (CRP).
* Demonstrate comprehension of the protocol procedures and knowledge of study by passing a written examination (passing grade is at least 80 percent).
* Capable of understanding, consenting and complying with the entire study protocol.
* Female subjects must be of non-childbearing potential, (as defined as surgically sterile or postmenopausal for more than 1 year), or if of childbearing potential must be practicing abstinence or using an effective licensed method of birth control (e.g., history of hysterectomy or tubal ligation; use hormonal or barrier birth control such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), cervical sponges, diaphragms, condoms with spermicidal agents, or must have a vasectomized partner) within 2 months of infection and must agree to continue such precautions during the study and for 30 days after the Day 56 study visit. Male subjects must agree not to father a child for 90 days after the Day 28 study visit. A woman is eligible if she is monogamous with a vasectomized male.
* Agrees not to participate in another clinical trial during the study period.

Exclusion Criteria:

* Women who are pregnant or lactating or have a positive serum pregnancy test at screening or positive urine pregnancy test upon admission to inpatient facility.
* Abnormal Vital signs, defined as:

  * Hypertension (systolic blood pressure >140 mm Hg or diastolic blood pressure >90 mm Hg) at rest on 2 separate days; or (heart rate <55 at rest on 2 separate days)
  * Respiratory rate >17
  * Temperature >/= 38.0 C (100.4 F) or symptoms of an acute self-limited illness such as an upper respiratory infection or gastroenteritis within 7 days of inoculum.
* Active positive Hepatitis B, C, and Human Immunodeficiency Virus (HIV) serologies.
* History of antimicrobial treatment in the 2 weeks before bacterial inoculum
* Received previous experimental E. coli, LT, or cholera vaccines or live E. coli or Vibrio cholerae challenges; or previous infection with cholera or diarrheagenic E. coli.
* Abnormal bowel habits as defined by fewer than 3 stools per week or more than 2 stools per day in the past 6 months.
* History of chronic gastrointestinal illness, including severe dyspepsia (mild or moderate heartburn or epigastric pain occurring no more than 3 times per week is permitted), lactose intolerance, or other significant gastrointestinal tract disease.
* Regular use (weekly or more often) of laxatives, anti-diarrheal, anti-constipation, or antacid therapy.
* History of major gastrointestinal surgery, excluding uncomplicated appendectomy or cholecystectomy.
* Long-term use of oral steroids, parenteral steroids, or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (Nasal and topical steroids are allowed).
* Have a diagnosis of schizophrenia or other major psychiatric diagnosis.
* Receiving the following psychiatric drugs: aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, molindone, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, chlorprothixene, chlorpromazine, perphenazine, trifluopromazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate
* History of receiving immunoglobulin or other blood product within the 3 months before enrollment in this study.
* Traveled to Enterotoxigenic Escherichia coli (ETEC) endemic areas within the past 2 years, ever having used Cholera/ETEC vaccine (Dukoral) or having been raised in a cholera or ETEC endemic area.
* Received any licensed vaccine within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) before enrollment in this study.
* An acute or chronic medical condition that, in the opinion of the investigator, would render ETEC infection unsafe or would interfere with the evaluation of responses. This includes, but is not limited to: known or suspected immunodeficiency, known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, history of diabetes, cancer (other than a healed skin lesion), heart disease (in the hospital for a heart attack, history of irregular heart beat or fainting caused by an irregular heart beat), unconsciousness (other than a single brief "concussion"), seizures (other than with fever when subject was a child <5 years old), asthma requiring treatment with inhaler or medication in the prior 2 years, autoimmune disease or eating disorder, and transplant recipients.
* Received an experimental agent (vaccine, drug, biologic, device, blood product or medication) within 1 month before enrollment in this study or expects to receive an experimental agent during the study.
* History of alcohol or drug abuse in the last 5 years.
* Planned to travel abroad in the time between vaccination and 30 days following the ETEC inoculum dose.
* Any condition that would, in the opinion of the Site Investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* Use of prescription and over-the-counter (OTC) medications that contain acetaminophen, aspirin, ibuprofen, and other nonsteroidal anti-inflammatory drugs within 48 hours prior to receiving the investigational product.
* Use of prescription acid suppression medication or OTC antacids within 72 hours of investigational product administration.
* Subjects with autoimmune disorders, chronic inflammatory disorders or neurological disorders with a potential autoimmune correlation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-12 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Diarrheal disease | 5 days
Adverse event monitoring | 30 days

SECONDARY OUTCOMES:
Immune responses towards challenge strain | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Halvor Sommerfelt, MD, PhD, Study Chair — Centre for International Health, University of Bergen
Locations (1):
- Haukeland University Hospital, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: Yes
Data and samples may be shared with current and future partners

REFERENCES:
- [Background] Skrede S, Steinsland H, Sommerfelt H, Aase A, Brandtzaeg P, Langeland N, Cox RJ, Saevik M, Wallevik M, Skutlaberg DH, Tellevik MG, Sack DA, Nataro JP, Guttormsen AB. Experimental infection of healthy volunteers with enterotoxigenic Escherichia coli wild-type strain TW10598 in a hospital ward. BMC Infect Dis. 2014 Sep 4;14:482. doi: 10.1186/1471-2334-14-482. PMID 25190096
- [Background] Aase A, Sommerfelt H, Petersen LB, Bolstad M, Cox RJ, Langeland N, Guttormsen AB, Steinsland H, Skrede S, Brandtzaeg P. Salivary IgA from the sublingual compartment as a novel noninvasive proxy for intestinal immune induction. Mucosal Immunol. 2016 Jul;9(4):884-93. doi: 10.1038/mi.2015.107. Epub 2015 Oct 28. PMID 26509875
- [Background] Sahl JW, Steinsland H, Redman JC, Angiuoli SV, Nataro JP, Sommerfelt H, Rasko DA. A comparative genomic analysis of diverse clonal types of enterotoxigenic Escherichia coli reveals pathovar-specific conservation. Infect Immun. 2011 Feb;79(2):950-60. doi: 10.1128/IAI.00932-10. Epub 2010 Nov 15. PMID 21078854
- [Background] Steinsland H, Lacher DW, Sommerfelt H, Whittam TS. Ancestral lineages of human enterotoxigenic Escherichia coli. J Clin Microbiol. 2010 Aug;48(8):2916-24. doi: 10.1128/JCM.02432-09. Epub 2010 Jun 9. PMID 20534806
- [Derived] Rim S, Sakkestad ST, Zhou F, Gullaksen SE, Skavland J, Chauhan SK, Steinsland H, Hanevik K. Dynamics of circulating lymphocytes responding to human experimental enterotoxigenic Escherichia coli infection. Eur J Immunol. 2023 Aug;53(8):e2250254. doi: 10.1002/eji.202250254. Epub 2023 Jun 28. PMID 37102399
- [Derived] Sakkestad ST, Steinsland H, Skrede S, Lillebo K, Skutlaberg DH, Guttormsen AB, Zavialov A, Paavilainen S, Soyland H, Saevik M, Heien AR, Tellevik MG, Barry E, Langeland N, Sommerfelt H, Hanevik K. A new human challenge model for testing heat-stable toxin-based vaccine candidates for enterotoxigenic Escherichia coli diarrhea - dose optimization, clinical outcomes, and CD4+ T cell responses. PLoS Negl Trop Dis. 2019 Oct 30;13(10):e0007823. doi: 10.1371/journal.pntd.0007823. eCollection 2019 Oct. PMID 31665141